CLINICAL TRIAL: NCT06051786
Title: An Open-label, Randomized, Parallel-Group, Multi-Site Study to Evaluate the Efficacy and Safety of Azelastine HCl-Fluticasone Propionate Nasal Spray 137-50 mcg/Spray in Perennial Allergic Rhinitis Patients
Brief Title: A Study to Evaluate the Safety and Effectiveness of a Nasal Spray to Treat Perennial Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Synmosa Biopharma Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFC-TW-001
Record Dates: First submitted 2023-08-31; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-08

CONDITIONS: Allergic Rhinitis
Keywords: Azelastine; Fluticasone
MeSH Terms: conditions — Rhinitis, Allergic | interventions — azelastine; Fluticasone; Nasal Sprays

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- azelastine hydrochloride and fluticasone propionate, 137/50 mcg (Experimental): The test product, azelastine hydrochloride and fluticasone propionate, 137/50 mcg is manufactured by the sponsor, administered as one spray in each nostril twice daily for 28 days.
  Interventions: Drug: azelastine/fluticasone 137/50 mcg nasal spray
- Dymista™ (Active Comparator): The active control product, Dymista™, is manufactured by Meda Pharmaceuticals, administered as one spray in each nostril twice daily for 28 days.
  Interventions: Drug: Dymista™

INTERVENTIONS:
Drug: azelastine/fluticasone 137/50 mcg nasal spray — AFC is a fixed-dose combination product of Azelastine hydrochloride (137mcg), a selective H1-receptor antagonist and, Fluticasone propionate (50mcg), a corticosteroid. AFC is administered intranasally and is used to treat Allergic Rhinitis (AR).
  Other Names: AFC
  Arms: azelastine hydrochloride and fluticasone propionate, 137/50 mcg
Drug: Dymista™ — Dymista™ is a fixed-dose combination product of Azelastine hydrochloride (137mcg), a selective H1-receptor antagonist and, Fluticasone propionate (50mcg), a corticosteroid. Dymista™ is administered intranasally and is used to treat Allergic Rhinitis (AR).
  Other Names: AZE/FLU
  Arms: Dymista™

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Azelastine HCl-Fluticasone propionate Nasal Spray 137-50 mcg/spray compared to Dymista™ in patients with perennial allergic rhinitis

DETAILED DESCRIPTION:
This study is an open label, randomized, parallel-group study to evaluate the efficacy and safety of azelastine/fluticasone 137/50 mcg nasal spray, to Dymista™ nasal spray in perennial allergic rhinitis (PAR) patients.

An estimated 200 evaluable subjects are planned for this study. Subjects who are at least 20 years of age with PAR and meet the eligibility criteria will be eligible for this study.

There will be a 7-day washout period to establish a baseline, followed by a 28-day treatment period. All subjects who qualify after the washout period will be randomized to receive the test formulation of azelastine/fluticasone or Dymista™ during the treatment period, administered as one spray in each nostril twice daily for 28 days.

Subjects will self-score their symptoms twice daily (AM and PM, approximately 12 hours apart at the same times daily) throughout the washout period and the treatment period. During the treatment period, scoring should be made immediately prior to each dose to reflect the previous 12 hours (reflective scores). The 4 symptoms evaluated are: runny nose, sneezing, nasal itching, and congestion. Each of the symptoms will be scored on a scale of 0 to 3, with 0 indicating absent symptoms and 3 indicating severe symptoms (symptoms that are hard to tolerate; causes interference with activities of daily living and/or sleeping).

The primary endpoint is the difference in the mean change in reflective total nasal symptom scores (rTNSS) from baseline to the end of the treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. 20 years of age and older.
2. For female subjects of childbearing potential: agreement to practice birth control for the duration of the study with either A. A birth control form with a failure rate of < 1%: intrauterine device, hormonal contraceptive and abstinence; or B. A combination of birth control forms resulting in a failure rate of < 1%: male condom, female condom or diaphragm in combination with another adequate form of birth control (intrauterine device, hormonal contraceptive, male condom, female condom or diaphragm).
3. A medical history consistent with AR as judged by the investigator.
4. Allergy to perennial allergen demonstrated by Multiple Antigen Simultaneous Test (MAST) or ImmunoCAP test (> or = Class 1) within 12 months of the screening visit or during screening as assessed by the investigator.
5. If receiving immunotherapy injections, on a stable regimen for at least 30 days prior to Visit 2. Immunotherapy injections are defined as controlled repetitive dosing of allergen(s) at regular intervals, in order to increase immune tolerance to the offending allergen(s).
6. In order to enter the washout period, a reflective TNSS score of at least 6 on Visit 2.
7. In order to enter the treatment period, a Baseline reflective TNSS score of at least 6. The Baseline rTNSS is the mean of the rTNSS scores for the last 3 days of the washout period and the rTNSS score at the randomization visit.
8. Signed written informed consent.

Exclusion Criteria:

1. For females: Pregnancy, lactating, or planning to become pregnant during the study period.
2. Active or quiescent tuberculosis infections of the respiratory tract; Active and untreated local or systemic fungal, bacterial, viral, or parasitic infections within the 12months prior to the screening visit.
3. Presence of glaucoma, cataracts, ocular herpes simplex, conjunctivitis, or other eye infection within the 12 months prior to the screening visit.
4. Presence of any clinically significant nasal mucosal erosion, nasal septal ulcers, or septum perforation on focused nasal examination.
5. Nasal or sinus surgery or nasal trauma within the previous year likely to affect deposition of intranasal medication in the judgment of the investigator.
6. Other nasal disease(s) likely to affect deposition of intranasal medication, such as chronic sinusitis, rhinitis medicamentosa, clinically significant polyposis, or clinically significant nasal structural abnormalities (patients with severe nasal septum deviation, nasal stenosis or cleft lip and cleft palate).
7. Presence or history of any clinically significant condition that, in the judgment of the investigator, would compromise the safety of the subject or the conduct of the study.
8. Use of any investigational drug within 30 days prior to Visit 2.
9. Hypersensitivity to azelastine hydrochloride, fluticasone propionate, or any inactive ingredients of the investigational product.
10. Respiratory tract infection requiring antibiotics within 14 days prior to Visit 2.
11. Has clinically significant pulmonary disease, including asthma (with the exception of mild intermittent asthma) or chronic obstructive pulmonary disease (COPD).
12. Known history of alcohol, drug, or substance abuse in the 12 months prior to screening.
13. Use of any prohibited medications and treatments (including antihistamines, decongestants, leukotriene antagonists, corticosteroids and other nasal therapies,) within the time period specified in the protocol prior to Visit 2.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2021-07-20 (Actual)

PRIMARY OUTCOMES:
Change in reflective total nasal symptom scores (rTNSS) | 4 weeks
  Subjects will self-score their symptoms twice daily (AM and PM, approximately 12 hours apart at the same times daily) throughout the washout period and the treatment period. During the treatment period, scoring should be made immediately prior to each dose to reflect the previous 12 hours (reflective scores). The 4 symptoms evaluated are: runny nose, sneezing, nasal itching, and congestion. Each of the symptoms will be scored on a scale of 0 to 3, with 0 indicating absent symptoms and 3 indicating severe symptoms (symptoms that are hard to tolerate; causes interference with activities of daily living and/or sleeping).

SECONDARY OUTCOMES:
Nasal examinations | 4 weeks
  The Nasal Examination includes an evaluation for nasal irritation, epistaxis, and additional nasal symptoms including mucosal edema, nasal discharge, mucosal erythema, mucosal bleeding, and crusting of mucosa.
Adverse events | 4 weeks
  An adverse event is any untoward or unfavorable medical occurrence in a human subject, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the subject's participation in the research, whether or not considered related to the subject's participation in the research.

CONTACTS AND LOCATIONS:
Overall Officials: Te-Huei Yeh, MD, Principal Investigator — National Taiwan University Hospital
Locations (5):
- Taiwan (5):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Cathay General Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No